CLINICAL TRIAL: NCT03674697
Title: The Effect of Light Therapy on Post-Surgical Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Mohab Ibrahim, PhD MD, Associate Professor Anesthesiology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1808848766
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Acute Pain; Arthropathy of Knee
MeSH Terms: conditions — Acute Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Treatment Group (Green LED) (Experimental): Subjects will be exposed to a Green LED light for 8 weeks prior to surgery, during their hospital stay and for an additional 2 weeks after hospital discharge.
  Interventions: Device: Green LED light therapy
- Control Group (White LED) (Placebo Comparator): Subjects will be exposed to a White LED light for 8 weeks prior to surgery, during their hospital stay and for an additional 2 weeks after hospital discharge.
  Interventions: Device: White LED light therapy

INTERVENTIONS:
Device: Green LED light therapy — You will be asked to locate a dark room in your house 8 weeks prior to your surgery. You will place the provided LED strip near you on a flat surface and turn it on for 2 hours a day until the day of the surgery (8 weeks). You have the freedom to pick anytime during day or night to use the light. We will ask you to be as consistent as possible with your chosen time. You can engage in any activity to pass the time as long as it does not involve exposure to another light from an outside source (computers, TV, smartphones, tablets, etc.).
  Other Names: Treatment
  Arms: Active Treatment Group (Green LED)
Device: White LED light therapy — You will be asked to locate a dark room in your house 8 weeks prior to your surgery. You will place the provided LED strip near you on a flat surface and turn it on for 2 hours a day until the day of the surgery (8 weeks). You have the freedom to pick anytime during day or night to use the light. We will ask you to be as consistent as possible with your chosen time. You can engage in any activity to pass the time as long as it does not involve exposure to another light from an outside source (computers, TV, smartphones, tablets, etc.).
  Other Names: Control
  Arms: Control Group (White LED)

SUMMARY:
This is a prospective randomized clinical trial study to investigate two main aspects. The first aspect is to investigate the efficacy exposure to green light emitting diode (GLED) in reducing postoperative opioid medications requirements by 20% as the primary outcome amongst patients scheduled for elective total knee replacement surgery (knee arthroplasty). The second aspect is to reduce postoperative pain by 30%, improve preoperative anxiety by 30%, and improve the quality of sleep pre and postoperatively by 30%.

Seventy participants scheduled for elective unilateral primary total knee arthroplasty (total knee replacement) will be recruited from the pain clinic or from the orthopedic surgery clinics at Banner-University Medical Center by the pain or orthopedic physicians who are key personnel of this study. Once a participant is identified, he/she will meet with one of the research team members to explain the nature of the clinical trial and undergo a standard of care medical history gathering and baseline physical examinations. If the participant meets all the inclusion and have no exclusion criteria, he/she will be presented with a written consent in English to explain all the risk and benefits of this clinical trial. Once a participant signs a consent, he or she will be randomized by the study statistician, in a 1:1 ratio to either a GLED group (treatment) or white light-emitting diode (WLED) group (control). The participant will be trained on how to use the light device by one of the research team members. All participants will be exposed to either GLED or WLED for 8 weeks prior to surgery and two additional weeks after surgery.

DETAILED DESCRIPTION:
Participants who meet inclusion and exclusion criteria will be enrolled into the study after consenting. Patients will be interviewed and asked to provide their history of present conditions, past medical history, if they are on disability or receiving compensation for an injury, demographic information, and ethnic group (determined by self-identification). Additionally, patients will undergo a physical examination. The focus will be on the history of colorblindness and chronic pain. A pain assessment will be conducted, and this will be obtained verbally from the patient. Physical examinations will be obtained at the initial study visit and will be documented in the source documents.

The participants will be instructed to use the GLED or the WLED devices as follows:

Before surgery - The participants will be instructed to choose rooms in their home. These rooms must be dark and has no other source of light except the light device provided. The participants will be instructed to place the devices in their fields of vision and keep it between 3 feet away from their eyes. This distance is chosen based on the intensity of the light from our clinical trial, which corresponds to 100 lux. The participants will be asked not to stare directly at the light, but to rather allow it to enter their eyes from the periphery and to treat it as they would treat any other light fixture. The participants will be asked to have 2 hours of exposure every night. Given that participants may have different preferred time to go to bed, we will ask them to start the exposure any time after sunset when sunshine is no longer illuminating their chosen rooms for exposure. We will encourage the participants to participate in any activities that do not require additional lights so they do not fall asleep during the nightly light exposure. For example, the participants may enjoy reading (100 lux provide enough illumination for reading), listening to music, exercising, etc. The participants will be exposed nightly to their light for 8 weeks prior to surgery.

After Surgery - On average, half the participants may be discharged home from the hospital after they recover from anesthesia in the same day. The other half of the participants may be admitted to the hospital for 1-3 days on average based on their medical profile, the course of the surgery, and any complications or concerns of the surgeons or the anesthesiologists. For patients that will be discharged home on the same day, they will continue light exposure as they did before surgery. For patients who may be admitted to the hospital, we have already secured the approval from the hospital administrative staff as well as the nursing manager to allow the participants to utilize the light devices in the patients' rooms. The light devices were examined by the Facility Management (for electrical hazards) and Infection Control and both approved the use of the light devices in the hospital setting. The participants will place the light devices in their fields of vision in the patients' rooms. Patients and nurses are able to control the ambient lights in the rooms and it will be kept dark except for the light from the light devices for two hours every night. The participants will be exposed to the light for 2 hours in the evening prior to sleeping. If the surgery is scheduled late at night or if the participants has a slow emergence from anesthesia, they may not be awake during the first night in the hospital to have the light exposure. Once participants are discharged from the hospital, they will continue exposure to the light as they did before surgery for the remainder of the two weeks postoperatively.

Data Management:

Data will be collected on standardized case report forms and entered into a HIPPA-compliant electronic database (e.g. Microsoft Access) that provides an appropriate interface with a robust statistical package . All study-related hard copy materials will be stored in locked file cabinets.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years or older
2. Scheduled for elective primary knee replacement surgery
3. Able to understand, read, and write English

Exclusion Criteria:

1. History of chronic pain requiring chronic opioids equal or greater than 90 Morphine Milligram Equivalent (MME)/day
2. Severe psychological or psychiatric conditions
3. Unanticipated surgical complications, such as prolonged bleeding requiring long hospital stay, infection, dehiscence, and airway complications (anesthesiologist unable to extubate secondary to pulmonary complications
4. Surgery cannot be postponed eight weeks from the day of recruitment
5. Colorblindness
6. On disability, involved in a legal case pending, or receiving compensation for a work-related injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The amount of pain reducing medication used by the active treatment group and the control group. | 10 week period
  Change in postoperative opioid medications requirements by 20% as assessed by opioid medication logs

SECONDARY OUTCOMES:
The amount of pain reducing medication used by the active treatment group and the control group assessed by the Brief Pain Inventory survey. | 10 week period
  Change in postoperative pain by 30% as assessed by the Brief Pain Inventory survey
The amount of pain reducing medication used by the active treatment group and the control group assessed by Amsterdam Preoperative Anxiety and Information Scale survey. | 10 week period
  Change in preoperative anxiety by 30% as assessed by Amsterdam Preoperative Anxiety and Information Scale survey
The amount of pain reducing medication used by the active treatment group and the control group assessed by the Pittsburgh Sleep Quality Index survey. | 10 week period
  Change in the quality of sleep pre and postoperatively by 30% as assessed by the Pittsburgh Sleep Quality Index survey

CONTACTS AND LOCATIONS:
Overall Officials: Mohab Ibrahim, PhD, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hassett AL, Aquino JK, Ilgen MA. The risk of suicide mortality in chronic pain patients. Curr Pain Headache Rep. 2014;18(8):436. doi: 10.1007/s11916-014-0436-1. PMID 24952608
- [Result] Chau DL, Walker V, Pai L, Cho LM. Opiates and elderly: use and side effects. Clin Interv Aging. 2008;3(2):273-8. doi: 10.2147/cia.s1847. PMID 18686750
- [Result] Hwang MH, Shin JH, Kim KS, Yoo CM, Jo GE, Kim JH, Choi H. Low level light therapy modulates inflammatory mediators secreted by human annulus fibrosus cells during intervertebral disc degeneration in vitro. Photochem Photobiol. 2015 Mar-Apr;91(2):403-10. doi: 10.1111/php.12415. Epub 2015 Jan 26. PMID 25557915
- [Result] Ibrahim MM, Patwardhan A, Gilbraith KB, Moutal A, Yang X, Chew LA, Largent-Milnes T, Malan TP, Vanderah TW, Porreca F, Khanna R. Long-lasting antinociceptive effects of green light in acute and chronic pain in rats. Pain. 2017 Feb;158(2):347-360. doi: 10.1097/j.pain.0000000000000767. PMID 28092651